CLINICAL TRIAL: NCT07347704
Title: Evaluation of the Effectiveness of a Psychological Intervention for Fibromyalgia Supported by New Technologies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Collaborators: Hospital Provincial de Castellon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: FIBROEMA
Record Dates: First submitted 2021-10-28; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: We have included more participants than 20 because similar studies have recommended larger sample sizes for feasibility trials similar to ours
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Behavioral Therapy with app support (Experimental): A group intervention with a cognitive-behavioral approach of 8 sessions will be carried out. The intervention will focus on learning about the modulating factors of the pain experience and the acquisition of tools related to each of these factors.
  Interventions: Device: Cognitive Behavioral Therapy with app suport

INTERVENTIONS:
Device: Cognitive Behavioral Therapy with app suport — Psychotherapy based on Cognitive Behavioral Therapy principles supported with technology to receive notifications about the evolution of the participants during therapy

SUMMARY:
This study aims to evaluate the feasibility of a psychological intervention in patients diagnosed with Fibromyalgia supported by new technologies.

DETAILED DESCRIPTION:
Different therapeutic options for psychological intervention in fibromyalgia are currently available. However, these interventions are usually of a general nature and do not take into account the differences between patients.

On the other hand, we know that these programs have greater or lesser effectiveness in improving quality of life and adaptation to pain, but there is not as much information available regarding the therapeutic mechanisms that are related to this effectiveness, i.e., What variables mediate the improvement in therapy? When do they produce the change? Is it possible to adapt the interventions to the results of the same that we can receive in real time? In the present work we propose to apply a psychological treatment already validated for fibromyalgia emphasizing those variables of beliefs and coping that research has shown to be directly related to belonging to the group of higher or lower functionality.

The objective will be to find out, on the one hand, if it is feasible to monitor the change in therapy using new technologies and, on the other hand, to measure this change to consider it when implementing the intervention, which is traditionally quite manualized when performed at group level and hardly considers individual differences in the response to treatment during treatment. Specifically, by means of a validated App we will measure those therapeutic variables that we expect to change as a result of introducing the treatment and, if not, a series of alarms will be generated that will alert the clinician of the absence of the expected change so that he can adapt the intervention according to the evolution of the patient in real time.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with fibromyalgia

Exclusion Criteria:

* Does not have a smartphone

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
App' usability and acceptability | One administration one week after downloading the app
  The System Usability Scale will be used to evaluate the perception that this tool is simple to use and useful. It is composed by 10 items which are responded according to a 5-point Likert scale (1 = "completely disagree" to 5 ="completely agree").
Feasibility of the app | At the end of the study (9 weeks after study onset)
  Feasibility of the study will be assessed by a calculation of responses completed from the assessments prompted.

SECONDARY OUTCOMES:
Changes in the Fibromyalgia Impact Questionnaire | Changes from Pretreatment to Posttreatment (9 weeks after study onset)
  Evaluates impact of fibromyalgia on functioning. It includes 20 items with a response range from 0 to 10. Higher scores reflect greater impact of the disease.
Changes in the Chronic Pain Coping Inventory-42 | Changes from Pretreatment to Posttreatment (9 weeks after study onset)
  Evaluates coping strategies used to deal with pain. It includes 42 items scored from 0 days to 7 days depending on the number of days each coping strategy is used. Higher score means more frequent use of the strategy in the past week.
Changes in the Survey of Pain Attitudes | Changes from Pretreatment to Posttreatment (9 weeks after study onset)
  Evaluates beliefs about pain. It includes 25 items. Respondents are asked to indicate their degree of agreement using a 5-point Likert scale ranging from 0 (very false for me) to 4 (very true for me). A higher score on a subscale implies a greater degree of certainty about the corresponding belief or pain-related attitude.
Changes in the Beck Depression Inventory | Changes from Pretreatment to Posttreatment (9 weeks after study onset)
  Evaluates the severity of depression symptoms. It includes 21 items with a response range from 0 to 63. Higher scores reflect more severe depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Provincial, Castellon, Spain

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD